CLINICAL TRIAL: NCT04132791
Title: Chronotherapy With Aspirin for Reduction of Cardiovascular Disease
Brief Title: TIME ASPIRIN: Chronotherapy With Aspirin for Reduction of Cardiovascular Disease
Acronym: TImE ASPIRIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped prematurely due to too low inclusion rate
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, tnbonten, Assistant Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P18.127
Record Dates: First submitted 2019-06-07; First posted 2019-10-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases
Keywords: Aspirin; Chronotherapy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: parallel double blinded placebo controlled randomized clinical trial design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin after awakening + placebo before bedtime (Other): Acetylsalicylic acid 80 mg once daily, orally. Intake in de morning after awakening. Participants already use acetylsalicylic acid 80 mg once daily due to secondary prevention of cardiovascular disease.
  Placebo tablet once daily will be added to their medication. The placebo tablet will be taken before bedtime, orally. The placebo is given throughout the study.
  Interventions: Other: aspirin after awakening + placebo before bedtime
- placebo after awakening +aspirin before bedtime (Experimental): Acetylsalicylic acid 80 mg once daily, orally. The time will be changed form morning to bedtime. Participants already use acetylsalicylic acid 80 mg once daily due to secondary prevention of cardiovascular disease.
  Placebo tablet once daily will be added to their medication. The placebo tablet will be taken after awakening, orally. The placebo is given throughout the study.
  Interventions: Other: placebo after awakening + aspirin before bedtime

INTERVENTIONS:
Other: placebo after awakening + aspirin before bedtime — determine the difference in major adverse cardiovascular events between the group with aspirin after awakening and placebo before bedtime and the group with placebo after wakening and aspirin before bedtime.
  Other Names: Acetylsalicylic acid Cardio Teva 80 mg, intake before bedtime
  Arms: placebo after awakening +aspirin before bedtime
Other: aspirin after awakening + placebo before bedtime — determine the difference in major adverse cardiovascular events between the group with aspirin after awakening and placebo before bedtime and the group with placebo after wakening and aspirin before bedtime.
  Other Names: Acetylsalicylic acid Cardio Teva 80 mg, intake after awakening
  Arms: aspirin after awakening + placebo before bedtime

SUMMARY:
This study will be a comparative effectiveness research to determine the difference in major adverse cardiovascular events between the group with aspirin after awakening and placebo before bedtime and the group with placebo after awakening and aspirin before bedtime.

DETAILED DESCRIPTION:
Aspirin is the cornerstone of preventive cardiovascular disease (CVD) treatment and bedtime intake of aspirin (chronotherapy) has been shown to reduce morning activity of platelets. It has been shown that platelet reactivity follows a clear circadian rhythm, with a peak of platelet reactivity during the morning (6-12 AM). Importantly, studies have shown in meta-analyses that high platelet activity is predictive of adverse cardiovascular outcomes in patients with stable CVD. Given this knowledge, it is highly likely that the morning peak of platelet reactivity contributes to the morning peak of cardiovascular events and that reduction of morning platelet activity prevents cardiovascular events during morning hours. This may be achieved by intake of aspirin at bedtime instead of on awakening. This study will be a comparative effectiveness research to determine the difference in major adverse cardiovascular events between the group with aspirin after awakening and placebo before bedtime and the group with placebo after awakening and aspirin before bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Use of low-dose aspirin (acetylsalicylic acid 80mg [brand name: acetylsalicylic acid cardio TEVA]~)
* Patients using aspirin from an MDD ('Baxter')
* Capacity to give informed consent (IC)

Exclusion Criteria:

* Pregnancy
* Mental or physical disability to fulfil study requirements
* Insufficient knowledge of the Dutch language
* Patients currently participating in another (clinical) trial or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of major adverse cardiovascular events | maximum of 4 years follow up
  the difference in number of participants with a major adverse cardiovascular events, defined as the composite of death from cardiovascular causes, nonfatal myocardial infarction, or nonfatal stroke, transient ischemic attack, need for repeat revascularízation by redo-CABG or repeat percutaneous intervention.

SECONDARY OUTCOMES:
Comparing the incidence rate of major cardiovascular events between the two groups in the morning (6-12), evening (12-21) and night (21-6). | maximum of 4 years follow up
  It is expected that bedtime aspirin reduces the number of participants with primary outcome (major cardiovascular events) more during morning hours (6-12h) compared with the rest of the day. So we will compare the mornig events, afternoon/evening and night events between the two groups and compare the difference.
Incidence rate of side-effects between the 2 groups | maximum of 4 years follow up
  the difference between the 2 groups of the number of participants that experience side-effects (e.g. bleeding, gastrointestinal symptoms)
cost-effectiveness of the intervention | maximum of 4 years follow up
  Comparing the relative costs and outcomes (effects) between the 2 groups. Data from questionnaire (use of health care) and data from the primary and secondary health care systems. We can compare the use of health care between the two groups en we can calculate the difference in cost between the two groups. So we can estimate if our intervention is cost-effective.

OTHER OUTCOMES:
difference in quality of life | maximum of 4 years follow up
  Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level per dimensions can be coded as a number 1-5, which indicates having no problems for 1 and having extreme problems for 5. We can define 3,125 (=55) different health states. We compare the average health status of the groups at the beginning and at the end of the study. See if there is a difference in health status/ quaulity of life between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bonten, Principal Investigator — Leiden University
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided in our data management plan